CLINICAL TRIAL: NCT05723380
Title: Perfusion Index Value in Predicting the Clinical Outcome of Thoracic ESPB
Brief Title: Prediction of Clinical Outcome in Thoracic ESPB
Status: Completed | Type: Observational
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Other Study IDs: 2023-01-025-02
Record Dates: First submitted 2023-02-03; First posted 2023-02-10 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2023-02

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Erector spinae plane block — T2 ESPB group where ESPB is performed at T2 with local anesthetics 20ml

SUMMARY:
The primary endpoint of this study was to identify that Perfusion index (PI) has any predictive value for the treatment outcome of cervical radiculopathy

DETAILED DESCRIPTION:
The erector spinae plane block (ESPB) is a less invasive, safer, and technically easy alternative procedure to conventional neuraxial anesthetic techniques. In contrast to common neuraxial techniques such as paravertebral and epidural injections, the ESPB targets an interfascial plane which is far from the spinal cord, root, and pleura. First applied to thoracic neuropathic pain, currently ESPB is being applied to postoperative pain control and includes variable clinical situations. In the abdomen and thoracic wall, thoracic ESPB can be applied for pain control after cardiac surgery, video-assisted thoracic surgery, laparoscopic cholecystectomy, and thoracotomy. Recently, favorable postoperative pain control after lumbar spinal or lower limb surgeries has been reported with lumbar ESPB. In addition, ESPB has also been used for chronic pain conditions in the upper and lower extremities. The perfusion index (PI) is a numerical value for the ratio between pulsatile and non-pulsatile blood flow measured by a special pulse oximeter. Although the special probe for PI measurement is relatively more expensive compared with ordinary pulse oximetery probes, its benefit as a marker of peripheral perfusion and as an idex for sympathetic stimulation have increased its use progressively. PI has been used widely for the prediction of success of brachial plexus block or axillary block. Changes of PI ratio value showed an excellent predictive value for the success of block. There have been no studies demonstrating predictive value of PI in thoracic ESPB for the relief of cervical radiulopathy

ELIGIBILITY:
Inclusion Criteria:

* Cervical foraminal stenosis
* Cervical central stenosis
* Cerivcal disc herniation
* Cervical spondylolisthesis

Exclusion Criteria:

* infection
* pregnancy
* allergy to local anesthetic agents
* previous cervical spine surgery

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who visited the pain clinic
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Perfusion index changes among 4 time periods | baseline, 10 minutes after erector spinae plane block, 20 minutes after erector spinae plane block, 30 minutes after erector spinae plane block
  Perfusion index changes among 4 time periods
Number of patients showing numerical rating scale reduction more than 50% | 1 month after ESPB
  Number of patients showing numerical rating scale reduction more than 50%
Number of patients showing numerical rating scale reduction less than 50% | 1 month after ESPB
  Number of patients showing numerical rating scale reduction less than 50%
Number of patients showing no reduction in numerical rating scale | 1 month after ESPB
  Number of patients showing no reduction in numerical rating scale
Neck disability index changes between 2 time periods | baseline, 1 month after ESPB
  Neck disability index changes between 2 time periods

CONTACTS AND LOCATIONS:
Overall Officials: Ji H Hong, Principal Investigator — Keimyung University
Locations (1):
- Ji Hoon Park, Daegu, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No